CLINICAL TRIAL: NCT03580057
Title: Effect of Weight Loss and Lactation on Cardiovascular Risk Factors (the EVA-trial)
Brief Title: Effect of Weight Loss and Lactation (the EVA-trial)
Acronym: EVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Hilde Kristin Brekke, Professor, University of Oslo
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2017/FO148194
Record Dates: First submitted 2018-04-30; First posted 2018-07-09 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Risk Factor
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Breastfeeding promotion intervention (BPI) (Experimental)
  Interventions: Behavioral: Breastfeeding promotion intervention
- Diet- and weight loss intervention (D) (Experimental)
  Interventions: Behavioral: Diet and weight loss intervention
- BPI and D (Experimental): Both interventions.
  Interventions: Behavioral: Breastfeeding promotion intervention; Behavioral: Diet and weight loss intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Breastfeeding promotion intervention — Promotion (education, support and supervision) of breastfeeding by experienced breastfeeding consultants and midwife, in order to follow the Norwegian guideline of 6 months exclusive breastfeeding and partial breastfeeding for a year.
  Arms: BPI and D; Breastfeeding promotion intervention (BPI)
Behavioral: Diet and weight loss intervention — 12-week program of dietary behavior modification treatment (LEVA-method by Bertz et al. Am J Clin Nutr 2012;96:698), leading to 6 kg weight loss (0.5 kg per week) and a healthier diet (less sugar, snacks, full fat products, more vegetables and fruit, smaller portion sizes). Weight is monitored by phone contact every second week. After 12 weeks, the women are followed up by e-mail contact for 9 additional months.
  Arms: BPI and D; Diet- and weight loss intervention (D)

SUMMARY:
A randomized controlled trial aiming to investigate the effects and possible interactions of diet induced weight loss and lactation on cardiometabolic profile

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in gestational week <32, with a pre-pregnant BMI 25-35 kg/m2
* Residence in Oslo/Bærum and surrounding area
* Intention to breastfeed their child
* Able to read and write in Norwegian.

Exclusion Criteria:

* Medication that influences lipid or glucose metabolism
* Chronic disease that influences lipid or glucose metabolism (e.g. diabetes (World Health Organization, WHO, 2006) or diabetes in pregnancy (WHO 2013))
* Premature birth (before week 36)
* Preeclampsia
* Previous breast reducing surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only pregnant women are eligible
Enrollment: 156 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in body weight (kg) between visits. | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  Measured in light clothing without shoes. Together with measured height (m) will be used to calculate Body Mass Index.
Changes in markers of lipid- and glucose metabolism between visits. | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  Measured in mmol/l: total cholesterol, low-density lipoprotein, high-density lipoprotein, triglycerides and glucose In percentage: HbA1c In pmol/l: insulin.

SECONDARY OUTCOMES:
Changes in lipid subclasses (mmol/l), lipoprotein size (nm) and apolipoproteins between visits | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  In g/l: apolipoprotein (apo) B and apo A1. In mmol/l: lipoprotein (a)
Changes in blood pressure, diastolic and systolic between visits | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)
  Measured after 5 min rest, mean of last 2 of 3 measurements (mmHg)
Changes in waist and hip (cm) circumference between visits | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  A measuring tape specifically designed for waist circumference (Seca) will be used according to a standardized procedure Measurements will be taken against the skin at the approximate midpoint between the lower margin of the last palpable rib and the top of the iliac crest. Hip is measured over the widest point on the buttocks.
Changes in body composition (fat free mass in kg and fat mass in kg) between visits. | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  Measured by Bioelectrical impedance and Dual X-ray Absorptiometry

OTHER OUTCOMES:
Changes in circulating inflammation markers such as cytokines, high sensitivity C-Reactive Protein (hsCRP), CRP and microCRP between visits. | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  Measured in mg/l
Changes in environmental toxins in breast milk and blood, such as dioxines and Persistent Organic Pollutants (POPs) between visits. | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  Presented on lipid weight basis (ng/g)
Changes in plasma metabolomics such as lactate, pyruvate, citrate and amino acids between visits. | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  Measured in mmol/l
Changes in PBMC (peripheral blood mononuclear cell) gene expression levels of markers of inflammation and lipid metabolism between visits. | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  Changes in levels of markers of inflammation and lipid metabolism at PBMC gene expression level.
Changes in hemostatic markers such as plasminogen activator inhibitor-1 (PAI-1) antigen and von Willebrand factor (vWF) between visits. | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  PAI-1 measured in ng/mL, vWF measured in IU/dl
Changes in hormones such as prolactin, estradiol, progesterone between visits. | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  Measured in nmol/l
Changes in markers of micronutrient status such as Hb, ferritin and vitamin D between visits. | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  Ferritin will be evaluated in relation to CRP.
Changes in dietary intake (kcal) and nutrient composition measured by 4-day weighed diet record between 3 visits | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  Nutrient composition calculation in nutrient composition software Dietist Net Pro
Changes in physical activity (METs, activity counts, step counts) between visits. | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  measured by ActiGraph (GT3X)
Changes in quality of life (QOL) measured by RAND 36-Item Short-Form Health Survey Instrument (SF-36) between visits. | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  The SF-36 RAND consists of 36 questions grouped into 8 dimensions: physical functioning, limitations in physical role functioning, bodily pain, general health, vitality, social functioning, limitations in emotional role functioning, and mental health. Each dimension is scored from 0 (worst imaginable health) to 100 (best imaginable health).
Changes in quality of life (QOL) measured by EuroQol 5D (EQ-5D-5L) between visits. | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  EQ-5D-5L measures 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression (self-classified). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions (levels of perceived problems from 1. level indicating no problem to 5. level indicating extreme problems). This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state. EQ-5D-5L health states may be converted into a single index value.The index values, presented in country specific value sets, facilitates the calculation of quality-adjusted life years (QALYs) that will be used to inform economic evaluations of the interventions.
Changes in quality of life (QOL) measured by EuroQol Visual Analog Scale (EQ-VAS) between visits. | Visit 1 (2 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (post weaning ~15 months postpartum)
  The EQ-VAS records the respondent's self-rated health on a 20-cm visual analogue scale . The scale is numbered from 0 (the worst health you can imagine) to 100 (the best health you can imagine.) This information can be used as a quantitative measure of health.

CONTACTS AND LOCATIONS:
Overall Officials: Hilde K Brekke, PhD, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ohman EA, Fossli M, Rasmussen KM, Winkvist A, Loland BF, Holven KB, Brekke HK. Effects of Breastfeeding Promotion Intervention and Dietary Treatment in Postpartum Women with Overweight and Obesity: Results from a Randomized Controlled Trial on Weight and Cardiometabolic Risk Factors. J Nutr. 2024 Aug;154(8):2448-2458. doi: 10.1016/j.tjnut.2024.06.006. Epub 2024 Jun 18. PMID 38901636